CLINICAL TRIAL: NCT05233059
Title: The Feasibly, Efficacy, and Acceptability of FitEx for Endometrial Cancer Survivors: A Pilot Randomized Controlled Trial of Walking With or Without Yoga
Brief Title: FitEx for Endometrial Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-1256
Record Dates: First submitted 2021-08-02; First posted 2022-02-10 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Quality of Life; Cancer of Endometrium; Behavior, Health; Self Efficacy
Keywords: Walking; Yoga; Physical Activity Adherence; Goal Setting; Social Support
MeSH Terms: conditions — Endometrial Neoplasms; Health Behavior

STUDY DESIGN:
Intervention Model Description: 2 arm randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking (Active Comparator): The walking group will receive a tailored FitEx for endometrial cancer survivors, including cancer specific newsletters.
  Interventions: Behavioral: FitEx; Behavioral: Weekly Movement Sessions
- Walking Plus Yoga (Experimental): The walking group will receive a tailored FitEx for endometrial cancer survivors with yoga cuing and yoga-based newsletters.
  Interventions: Behavioral: FitEx; Behavioral: Weekly Yoga Sessions

INTERVENTIONS:
Behavioral: FitEx — FitEx is an 8 week goal-setting, behavior tracking, physical activity intervention with a low dose of social support which will be delivered virtually.
Behavioral: Weekly Yoga Sessions — 30 minutes of optional guided yoga online led by a 500 hour yoga teacher once a week for participants in the walking plus yoga arm. Also accompanied by a yoga based newsletter.
  Arms: Walking Plus Yoga
Behavioral: Weekly Movement Sessions — 30 minutes of optional guided movement online led by a 500 hour yoga teacher once a week for participants in the walking arm. Also accompanied by a movement based newsletter.
  Arms: Walking

SUMMARY:
The purpose of this study is to determine whether a physical activity tracking program called FitEx would be useful to endometrial cancer survivors. Each interested endometrial cancer survivor will recruit 1 to 5 additional friends/family members to participate in the intervention with them, forming a team.

Each team will be randomized to FitExEC (control group) that receives FitEx for endometrial cancer survivors, or FitExEC+yoga (experimental group) that receives FitEx for endometrial cancer survivors plus yoga cueing. FitExEC is based on FitEx, a program used to encourage adults to improve their fruit and vegetable intake while increasing their physical activity. FitEx works by having participants join a team with their friends and loved ones, so they can support one another in meeting their goals. In this study, teams of endometrial cancer survivors/support members will receive watches that track how much they walk.

Each day, participants record how much exercise, how many fruits, and how many vegetables they've eaten that day for a total of 8 weeks. Participants will be encouraged to attend a virtual session 15 minutes per week that will focus on 1-mile worth of exercise points (all control) or 15 minutes of yoga (all experimental) followed by 15 minutes of support (endometrial cancer survivors only [control and experimental survivors in different groups]).

Participation in the study lasts roughly 10 weeks, and participants will be followed for 6 months afterward. The investigators think that FitEx may help people with endometrial cancer improve their daily physical activity and slowly improve their health and quality of life. The investigators hypothesize this intervention is feasible and acceptable to Carilion Clinic endometrial cancer survivors.

DETAILED DESCRIPTION:
Uterine cancer is the leading form of gynecologic malignancy in the United States. Currently, there are more than 600,000 EC survivors in the United States, and that number is expected to grow. Endometrial cancer (EC) is caused by excess estrogen, which acts as an oncogenic signal. Postmenopausal women with obesity have increased production of estrogen and are at an increased risk of developing type I EC.

Endometrial cancer was one of the first types of cancer to have an established relationship with body mass index (BMI). This relationship is linear and dose-dependent with BMI and can be explained by excess estrogen production . In women, adipose tissue is able to generate a form of estrogen known as estrone. Excess adipose tissue leads to increased production of estrone, which proliferates endometrial growth. For every five unit increase of BMI, the production of excess estrogen drives a 50% increased relative risk of developing EC.

Approximately 62% of American women are overweight or obese, putting them at increased risk of developing EC, the sixth most common cancer type in women in the United States. As the obesity rate in America continues to rise, the incidence of EC cases follows similar patterns. Between 2003 to 2015, the number of new EC diagnoses has increased by 13%, and continues to increase by 1% in following years. The National Cancer Institute predicts that nearly 60,000 new cases of EC will be diagnosed in 2021 and estimates that nearly 3% of women will be diagnosed with EC in their lifetime.

Fortunately, EC patients have relatively strong outcomes compared to other cancer types, as patients have an approximately 80% 5-year survival rate. However, a vast majority (70 - 90%) of type 1 EC survivors are obese. Five years after diagnosis, women with EC are more likely to die from cardiovascular disease and its risk factors, such as obesity and type 2 diabetes, than from EC. EC survivors with obesity report higher rates of depression and lower quality of life outcomes (sleep quality, self-esteem, fatigue, daily stress, etc.) than their non-obese counterparts. These outcomes worsen as BMI increases.

Addressing the role of obesity in EC survivors by encouraging physical activity is critical to improving optimal longitudinal care to survivors suffering from declining quality of life. Regular physical activity is associated with decreased levels of circulating estrogens in post-menopausal women and moderate physical activity in adulthood has been associated with reduced rates of developing endometrial cancer. As measured by a meta-analysis of physical activity interventions in participants with cancer, physical activity has established improvements to quality of life, fatigue, and physical functioning.

The connection between physical activity and BMI, morbidity, mortality, and improved quality of life outcomes is well supported. Despite this connection, only 1% of EC survivors meet all of the American Cancer Society guidelines for diet, exercise, and smoking recommendations. To increase the number of EC survivors meeting these guidelines, various exercise interventions have been developed to encourage EC survivors to increase physical activity and ultimately, improve their BMI.

However, existing interventions for EC survivors, geared towards improvements in BMI, have not been found to be efficacious in eliciting long-term changes in behavior with respect to weight loss. Because targeting weight loss was not effective in prior interventions, a successful intervention should target increasing physical activity rather than explicitly decreasing BMI. In breast cancer survivors, a similar demographic, many existing physical activity interventions are unsuccessful due to their focus on high intensity activities and due to the burden on participants to exercise together in person. In order to address pitfalls in prior physical activity studies, an ideal intervention should also target improvements to physical activity using lighter, ergonomically sound movements in a remote setting.

While participants report in-person physical activity as a barrier, various exercise studies have demonstrated that increasing social support is a powerful motivator of long-term behavior change, including adherence to physical activity. EC survivors surveyed in Canada report wanting a program that incorporates social support into an intervention. In breast cancer survivors, a group-dynamics based intervention achieved improvements in physical activity outcomes that persisted six months post-intervention.

Prior successful interventions have utilized social support but often require substantial physician engagement. While patients are more likely to engage with an exercise intervention if encouraged by their physician, oncologists noted barriers to promoting healthy behaviors in patients with obesity include lack of training in health promotion and even fear of overwhelming patients with health-promoting advice. Past ECS research that has shown successful and lasting improvements to behavior include weekly 1-on-1 physician calls and personalized telehealth communication, and cancer center exercise classes. In these interventions, an implicit cost is associated with staffing or availability (both for the participant and for the intervention facilitator). Taken together, an intervention that can facilitate the sense of groupness and be delivered virtually is optimal due to budget constraints on healthcare centers, geographical constraints of participants, and the current COVID-19 pandemic.

Surveyed EC survivors prefer gentle, group-based, walking exercises that function as support groups and exercises that they can do from home, but note barriers to adherence include access, fatigue, and pain. Yoga has been shown to decrease cancer-related fatigue, improve mobility, and increase mindfulness among cancer patients. Weekly yoga is a potential target to address barriers of exercise but has not been explored in detail in the EC patient population. In a focus group of sixteen gynecologic cancer survivors, yoga was viewed favorably by survivors and is a newly developing target for increased physical and psychological well-being. Yoga improvements have been shown in a range of health conditions including post-menopausal symptoms, cancer, heart disease, and even long-term improvements to BMI. The most common demographic for yoga practitioners is White, middle-aged women and practitioners strongly endorse the benefits of yoga on mindfulness, social support, and coping with stress. Prior work in EC survivorship has demonstrated that increased BMI has a negative impact on quality of life, an outcome that yoga has improved in similar populations such as breast cancer survivors.

Goal setting and behavior tracking are two key behavioral psychology principles that encourage and promote improvements in exercise and dietary habits in obese adults, and successful interventions should incorporate these principles as components to see greater success. FitEx is a virtual, scalable, evidence-based walking program that can be easily modified to include other exercises such as yoga. FitEx has shown significant maintenance of physical activity changes six months post-intervention. FitEx participants join a team, led by regional facilitators and local team captains, and set a physical activity and dietary goals throughout the eight week intervention. Participants have the opportunity to meet with others weekly for remote, guided exercise demonstrations. Participants are able to see if their goals are being met each week as self-monitoring is built into the FitEx interface, creating a sense of real time feedback. The program was developed for community-dwelling adults and its impact on cancer survivors has yet to be tested. Thus, FitEx is an intervention that meets the five dimensions of RE-AIM: Reach, Effectiveness, Adoption, Implementation, and Maintenance, such that small changes to FitEx do not diminish any of these dimensions and overall program success. Because FitEx is a validated program of measuring daily physical activity adherence which incorporates a low-dose of social support, it can easily be modified to target specific populations. Additionally, FitEx can be modified to include different exercises, such as yoga, which are viewed favorably by ECS. The present study seeks to determine whether a modified FitEx intervention geared towards survivorship or yoga improves outcomes in physical activity adherence and in quality of life in EC survivors.

As measured through FitEx, the yoga intervention will provide a remote workout regimen led by a registered yoga instructor. The control FitEx condition will include standard weekly meetings that currently take place in FitEx. Both arms incorporate walking as the predominant form of exercise and may include any other exercises of the participant's preference according to their goals. As a modified, tailored intervention for ECS, FitEx has the potential to improve physical activity adherence and quality of life in ECS.

The overall objective of this work is to tailor FitEx for ECS, with the goal of improving physical activity, as measured by step count, for both groups. Participants will be randomized to EC- tailored FitExEc (control) or FitExEC+yoga (intervention). The study hypotheses are (1) FitExEC and FitExEC+ yoga are feasible and acceptable (2) participants in both conditions will have improved weekly step count compared to baseline and (3) participants in the yoga-tailored condition will have greater improvements in quality of life compared to the ECS control condition.

The study's primary aims are feasibility and acceptability. The investigators will assess using recruitment statistics.

The study's secondary aims are efficacy related to physical activity improvement (measured through pedometers (step count) and subjectively through self report) as well as quality of life, fear of cancer recurrence, exercise preferences, social support, self-compassion, and exercise class satisfaction.

The investigators expect that both group-based programs will improve physical activity behaviors during the 8- week intervention, while the yoga-tailored group will exhibit improved secondary outcomes. The study's complementary aims will assess psychosocial factors, long-term outcomes, and barriers to implementation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with early stage (I-II) endometrial cancer, any histology
* Received cancer care at Carilion Clinic after 1/1/2010
* At least 18 years of age
* Have adequate comprehension (reading and writing) of the English language
* Have a BMI ≥ 30 kg/m^2 at screening
* Have stable internet access or access to a smartphone with internet
* Meet the requirements of the Physical Activity Readiness Questionnaire (PARQ)
* Have the capacity to provide informed consent and are willing to provide informed consent

Exclusion Criteria:

* History of recurrent endometrial cancer TARGET - Vital status: deceased
* Are meeting physical activity guidelines set forth by the American Cancer Society at screening (greater than 150 minutes/week of moderate physical activity, or greater than 75 minutes/week of vigorous physical activity)
* Have functional limitations requiring a walker, wheelchair, scooter, or other walking aid which limits their capacity to engage in the intervention safely

Healthy volunteers can be either gender with criteria below:

Inclusion Criteria:

* Were identified by a participant with endometrial cancer as a member of their support system
* Are at least 18 years of age
* Have adequate comprehension (reading and writing) of the English language
* Have stable internet access or access to a smartphone with internet capabilities
* Meet the requirements of the Physical Activity Readiness Questionnaire(PARQ)
* Have the capacity to provide informed consent and are willing to provide informed consent

Exclusion Criteria:

* Have functional limitations requiring a walker, wheelchair, scooter, or 6 other walking aid which limits their capacity to engage in the intervention safely

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Feasibility and Acceptability as measured by recruitment rate and program completion | 8 weeks
  Our primary aims are program adherence, measured as the percentage of participants who complete the 8 week program, and recruitment rate, measured as the percentage of participants who join the study out of the total participants who are approached about the study. These outcomes will be used to assess the feasibility and acceptability of the study among participants who enroll in the study and percentage of participants who complete the program.

SECONDARY OUTCOMES:
Changes to self-reported physical activity levels as measured by L-Cat questionnaire | 6 months
  The program surveys participants using the Stanford Leisure-Time Activity Categorical Item questionnaire pre and post-program to assess any changes to self-reported physical activity levels.
Changes to Quality of Life as measured by FACT-En questionnaire | 6 months
  The program will evaluate changes to quality of life, measured by pre and post program questionnaire (Functional Assessment of Cancer Therapy - Endometrial).
Changes to Yoga Self-Efficacy as measured by Yoga Self Efficacy questionnaire | 6 months
  The program will evaluate changes to yoga self efficacy as measured by the Birdee Yoga Self-Efficacy Scale at pre and post-program to determine whether this questionnaire is useful for future iterations of the study.
Self reported physical activity measured via steps per day on pedometer | 6 months
  We will assess participant's self reported daily step count, measured as total steps per day via pedometer.
Changes to Fear of Cancer Recurrence measured by Fear of Cancer Recurrence Inventory questionnaire | 6 months
  The program will evaluate changes to self-reported fear of cancer recurrence inventory as measured by fear of cancer recurrence inventory at pre and post-program to determine whether this questionnaire is useful for future iterations of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Armbruster, MD, MPH, Principal Investigator — Carilion Clinic Physician
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agnew H, Kitson S, Crosbie EJ. Interventions for weight reduction in obesity to improve survival in women with endometrial cancer. Cochrane Database Syst Rev. 2023 Mar 27;3(3):CD012513. doi: 10.1002/14651858.CD012513.pub3. PMID 36971688
- See also: Implementation Science — https://doi.org/10.1186/s13012-017-0640-6
- See also: Lancet — https://doi.org/10.1016/S0140-6736(05)67063-8
- See also: Complementary Therapies in Medicine — https://doi.org/10.1016/j.ctim.2014.12.003
- See also: PeerJ — https://doi.org/10.7717/peerj.3150
- See also: Gynecologic Oncology — https://doi.org/10.1016/j.ygyno.2014.01.025
- See also: American Psychological Association — https://www.apa.org/pubs/journals/hea
- See also: The Journal of Steroid Biochemistry and Molecular Biology — https://doi.org/10.1016/j.jsbmb.2013.05.001
- See also: Nature Reviews Cancer — https://doi.org/10.1038/nrc1408
- See also: Cancer of the Endometrium - Cancer Stat Facts — https://seer.cancer.gov/statfacts/html/corp.html
- See also: American Journal of Preventive Medicine — https://doi.org/10.1016/j.amepre.2016.05.011
- See also: Breast Cancer Research and Treatment — https://doi.org/10.1007/s10549-019-05278-w
- See also: Gynecologic Oncology — https://doi.org/10.1016/j.ygyno.2009.03.039
- See also: Complementary Therapies in Clinical Practice — https://doi.org/10.1016/j.ctcp.2010.09.007
- See also: FitEx — https://www.parcilab.org/fitex
- See also: British Journal of Sports Medicine — https://doi.org/10.1136/bjsports-2015-094787
- See also: Frontiers in Public Health — https://doi.org/10.3389/fpubh.2019.00064
- See also: Medicine and Science in Sports and Exercise — https://doi.org/10.1249/MSS.0000000000000360
- See also: Journal of Nutrition Education and Behavior — https://doi.org/10.1016/j.jneb.2018.12.010
- See also: Frontiers in Public Health — https://doi.org/10.3389/fpubh.2018.00071
- See also: JMIR MHealth and UHealth — https://doi.org/10.2196/mhealth.9563
- See also: International Journal of Behavioral Nutrition and Physical Activity — https://doi.org/10.1186/1479-5868-4-21
- See also: Key Statistics for Endometrial Cancer — https://www.cancer.org/cancer/endometrial-cancer/about/key-statistics.html
- See also: International Journal of Obesity — https://doi.org/10.1038/ijo.2013.36
- See also: Cochrane Database of Systematic Reviews — https://pubmed.ncbi.nlm.nih.gov/29388687/
- See also: BMJ Open — https://doi.org/10.1136/bmjopen-2017-018015
- See also: Oncology Nursing Forum — https://doi.org/10.1188/19.ONF.185-197
- See also: Supportive Care in Cancer: Official Journal of the Multinational Association of Supportive Care in Cancer — https://doi.org/10.1007/s00520-010-1066-8
- See also: American Journal of Obstetrics and Gynecology — https://doi.org/10.1016/0002-9378(78)90287-9
- See also: Journal of Behavioral Medicine — https://doi.org/10.1007/BF00844757
- See also: Gynecologic Oncology — https://doi.org/10.1016/j.ygyno.2013.12.023
- See also: Mindfulness — https://doi.org/10.1007/s12671-015-0479-3
- See also: Journal of Behavioral Medicine — https://doi.org/10.1007/s10865-015-9618-5
- See also: Complementary Therapies in Medicine — https://doi.org/10.1016/j.ctim.2014.08.008
- See also: The Journal of Steroid Biochemistry and Molecular Biology — https://doi.org/10.1016/S0960-0760(00)00113-8
- See also: Gynecologic Oncology — https://doi.org/10.1016/0090-8258(86)90103-4
- See also: RE-AIM - Reach Effectiveness Adoption Implementation Maintenance — https://www.re-aim.org
- See also: Hormones and Cancer — https://doi.org/10.1007/s12672-019-0358-9
- See also: Gynecologic Oncology — https://doi.org/10.1016/j.ygyno.2018.04.560
- See also: Journal of Gynecologic Oncology — https://doi.org/10.3802/jgo.2015.26.2.141
- See also: Preventive Medicine — https://doi.org/10.1016/0091-7435(87)90022-3
- See also: International Journal of Behavioral Nutrition and Physical Activity — https://doi.org/10.1186/s12966-017-0494-y
- See also: American Journal of Obstetrics and Gynecology — https://doi.org/10.1016/j.ajog.2011.05.042
- See also: Gynecologic Oncology — https://doi.org/10.1016/j.ygyno.2015.10.020
- See also: The International Journal of Behavioral Nutrition and Physical Activity — https://doi.org/10.1186/s12966-019-0789-2
- See also: International Journal of Behavioral Nutrition and Physical Activity — https://doi.org/10.1186/1479-5868-4-4
- See also: BMC Medicine — https://doi.org/10.1186/s12916-015-0323-6
- See also: BMC Geriatrics — https://doi.org/10.1186/s12877-017-0520-6
- See also: Uterine Cancer - Statistics — https://www.cancer.net/cancer-types/uterine-cancer/statistics
- See also: American Journal of Obstetrics and Gynecology — https://doi.org/10.1016/j.ajog.2005.03.038
- See also: Obstetrics & Gynecology — https://doi.org/10.1097/AOG.0b013e31820205b3
- See also: Gynecologic Oncology — https://doi.org/10.1016/j.ygyno.2012.04.013
- See also: Supportive Care in Cancer — https://doi.org/10.1007/s00520-020-05794-2
- See also: Journal of Molecular Endocrinology — https://doi.org/10.1530/JME-15-0310

DOCUMENTS (1):
  • Informed Consent Form (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT05233059/ICF_000.pdf